CLINICAL TRIAL: NCT01011452
Title: Assessment of the Effect of Oral Montelukast as Additional Treatment in the Management of Patients With Acute Severe Asthma.
Brief Title: Acute Montelukast in Asthma
Acronym: AcMk
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of East Anglia (Other)
Collaborators: Norfolk Association of Asthma Nurses (Unknown); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Crichton Ramsay, NNUH
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LREC 2000-108
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2009-11-11 (Estimated); Status verified 2009-11

CONDITIONS: Acute Asthma Exacerbation
Keywords: Acute Asthma Exacerbation; Montelukast; Management of acute asthma exacerbation
MeSH Terms: interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Montelukast (Active Comparator): 1 study capsule at study entry Montelukast 10mg and a further study capsule at 10pm for four weeks
  Interventions: Drug: Montelukast
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Montelukast — 1 study capsule at study entry Montelukast 10mg and a further study capsule at 10pm for four weeks
  Other Names: Singulair
  Arms: Montelukast
Drug: Placebo — 1 placebo capsule at study entry and a further placebo capsule at 10pm for four weeks
  Arms: Placebo

SUMMARY:
Patients presenting to hospital with an acute asthma exacerbation severe enough to require admission would receive full standard treatment according to British Thoracic Society guidelines in addition they would be offered the opportunity to take part in the study which would requite them to take a capsule of either montelukast or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Acute Asthma exacerbation requiring hospitalisation

Exclusion Criteria:

* Smoking history greater than or equal to 10 pack years
* Presenting PEFR greater than or equal to 75% predicted / best
* Failure to demonstrate greater than or equal to 15% variability in PEFR or FEV during the study
* Any significant and active pulmonary pathology other than asthma
* Pregnancy or breastfeeding
* Intended pregnancy or inability to take adequate precautions against conception
* Patient already on Montelukast
* Patient already on Phenobarbitone
* Patient already on Rifampicin
* Patient already on Phenytoin
* Chronic airflow limitation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2001-05; Primary Completion 2004-08 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Difference in peak flow between active and placebo limbs by the morning after randomization | 24 hours maximum

SECONDARY OUTCOMES:
Time (hours) to achieve PEF and FEV greater than or equal to 75% best achieved in the last 12 months with greater than or equal to 25% diurnal variation | 24 hours maximum
Time to discharge from hospital
PEF, FEV and FVC (as % best/predicted) the morning following admission and at 4 week clinic follow up
Proportion of days (post discharge until follow up) with a PEFR of less than or equal to 75%, and less than or equal to 50% best predicted
Proportion of days (post discharge until follow up) with a PEFR variability of greater than or equal to 25%
Residual volume as % predicted and RV/TLC% and FEF50 and FEF75 at 4 week out patient visit
requirement for further medical intervention / increases in treatment following discharge
Evaluation of quality of life over the four week out patient follow up period and expressed preference to continue on study medication
Evaluation of economic costs and savings from the additional treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Norfolk and Norwich University Hospital, Norwich, United Kingdom

REFERENCES:
- [Result] Ramsay, CF., Oral Motelukast in Patients with Acute Severe Asthma. Abstract NO P3609. ERJ Sept 2007
- [Derived] Ramsay CF, Pearson D, Mildenhall S, Wilson AM. Oral montelukast in acute asthma exacerbations: a randomised, double-blind, placebo-controlled trial. Thorax. 2011 Jan;66(1):7-11. doi: 10.1136/thx.2010.135038. Epub 2010 Oct 18. PMID 20956393